CLINICAL TRIAL: NCT06717074
Title: A Randomized, Double-blind, Placebo-controlled Phase IIa Trial to Evaluate Safety, Pharmacokinetics and Pharmacodynamics of Repeated Subcutaneously Administered RBD4059 in Participants With Stable Coronary Artery Disease
Brief Title: A Study to Evaluate Safety, Pharmacokinetics and Pharmacodynamics of RBD4059 in Participants With Stable Coronary Artery Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ribocure Pharmaceuticals AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC03T001
Record Dates: First submitted 2024-11-04; First posted 2024-12-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Stable Coronary Artery Disease CAD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low dose group, active (Experimental): Participants will receive RBD4059 as subcutaneous injections
  Interventions: Drug: RBD4059
- Low dose group, placebo (Placebo Comparator): Participants will receive placebo as subcutaneous injections
  Interventions: Drug: Placebo
- High dose group, active (Experimental): Participants will receive RBD4059 as subcutaneous injections
  Interventions: Drug: RBD4059
- High dose group, placebo (Placebo Comparator): Participants will receive placebo as subcutaneous injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RBD4059 — RBD4059, active drug.
  Arms: High dose group, active; Low dose group, active
Drug: Placebo — Placebo that is identical in appearance and volume to the doses of active IMP.
  Arms: High dose group, placebo; Low dose group, placebo

SUMMARY:
The goal of this clinical trial is to learn about the safety of drug RBD4059, and also if drug RBD4059 works to treat stable coronary artery disease in adults.

The main questions the trial aim to answer are:

What medical problems may participants experience when taking drug RBD4059? Researchers will compare drug RBD4059 to a placebo to see if drug RBD4059 works to treat stable coronary artery disease.

Participants will:

Receive drug RBD4059 or a placebo. Visit the clinic 11 or 12 times during 11 or 14 months for checkups and tests, depending on which treatment group they belong to.

DETAILED DESCRIPTION:
Low-dose group The trial will start with the low-dose group. The screening period takes place between D-28 to D-1 including informed consent, and those who meet the inclusion criteria and not meet any exclusion criteria will return to the trial site for further evaluating at D1 to confirm enrolment in the trial.

Participants will be assigned and randomized to receive RBD4059 (n=10) or placebo (n=5). All participants will be dosed at the trial site and undergo blood sampling and examinations at pre-defined timepoints.

A SRC meeting will be conducted on data from day 36 (W5), including at least 9 participants in the low-dose group. Provided acceptable safety profile of the low dose group, data from this SRC meeting will be used to guide initiation of the high-dose group.

Participants will return to the site and be monitored for safety and efficacy throughout the trial. Safety will be monitored until D336 (Week 48).

High-dose group This group will be initiated when the 36-day SRC meeting of the low-dose dose cohort has been conducted with no significant safety issues established. For the high-dose group, the screening period takes place between D-28 to D-1 including informed consent, and those who meet the inclusion criteria and not meet any exclusion criteria will return to the trial site for further evaluating at D1 to confirm enrolment in the trial.

Participants will be assigned and randomized to receive RBD4059 (n=10) or placebo (n=5). All participants will be dosed at the trial site and undergo blood sampling at pre-defined timepoints.

Participants will return to the site and be monitored for safety and efficacy throughout the trial until D426 (Week 60).

In both treatment groups, a switch from treatment with aspirin 75 mg to the equivalent AMP (Trombyl 75 mg) will be initiated on D1 and continue to the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the trial.
* Male or female (post-menopausal) participants ≥50-75 years.
* Patients with stable CAD defined as chronic coronary syndromes according to ESCs guideline on chronic coronary syndromes including the category asymptomatic or symptomatic patients more than 1 year after initial diagnosis or revascularization.
* Ongoing standard treatment with aspirin 75 mg for at least 3 months
* Stable prescription drugs i.e., ongoing since at least 30 days prior to randomization, should continue during the trial.

Main exclusion Criteria:

* Presence of any significant arrythmia in opinion of the investigator
* Any clinical suspicion on acute coronary syndrome or unstable angina at enrolment according to ESC criteria : (i) rest angina, i.e. pain of characteristic nature and location occurring at rest and for prolonged periods (more than 20 min); (ii) new-onset angina, i.e. recent (2 months) onset of moderate-to-severe angina (Canadian Cardiovascular Society grade II or III); or (iii) crescendo angina, i.e. previous angina, which progressively increases in severity and intensity, and at a lower threshold, over a short period of time.
* Patients with other clinical scenarios qualifying in the ESC definition of chronic coronary syndromes: patients with suspected CAD and 'stable' anginal symptoms, and/or dyspnoea, with new onset of heart failure (HF) or left ventricular (LV) dysfunction and suspected CAD, with angina and suspected vasospastic or microvascular disease.
* High bleeding risk defined as history of any significant bleeding (included but not limited to intracerebral haemorrhage and gastrointestinal), anaemia, liver failure, age more than 75 years or Clinical Frailty Score more than 5, or weight less than 60kg.
* Major surgery during last 30 days or planned major surgery or intervention within trial period.
* Capillary Hb less than 120 g/l for women and less than 130 g/L for men.
* Elective PCIor CABG within the previous 12 months.
* Previously confirmed ischemic stroke.
* Ongoing indication for chronic anti-coagulation therapy (incl. but not limited to patients with: atrial fibrillation, venous thrombo-embolism, mechanical cardiac valves) with NOACs, warfarin or other similar anticoagulants.
* Left ventricular ejection fraction (LVEF) less than 30% at enrolment.
* New York Heart Association (NYHA) class III-IV heart failure at entry, hospitalization for exacerbation of chronic heart failure within the previous 12 months or other indices of unstable heart failure.
* Creatinine clearance calculated by Cockcroft Gault equation less than 60ml/min*m2 at the time of enrolment. Hemodynamically significant valvular disease or valvular disease likely to require surgery within 3 years.
* Hemodynamically significant valvular disease or valvular disease likely to require surgery within 3 years.
* Expected survival time is less than one year for non-cardiac related disorders.
* History or presence of:

  1. Bleeding disorder(s) and/or at risk of bleeding, including relevant familial history.
  2. Thromboembolic diseases.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency, intensity and seriousness of reported AEs, SAEs and AEs of special interest (AESIs) during the trial. | From baseline until end of trial at week 48 or 60, depending on the dose group.
  Number and percentage of participants with AEs, SAEs and AEs of interest. All reported AE terms will be coded using Medical Dictionary for Drug Regulatory Affairs (MedDRA).

SECONDARY OUTCOMES:
Plasma concentrations of RBD4059. | In conjunction of administration of the IMP
Change and percent change compared with pre-dose baseline of FXI activity at different time points in each group. | From baseline until end of trial at week 48 or 60, depending on the dose group.
Proportion of participants with positive immunogenicity, measured as plasma concentrations of anti-drug antibodies (ADAs) | From randomization until end of trial at week 48 or 60, depending on the dose group.
Change and percent change compared with pre-dose baseline of APTT and PK(INR) at different time points in each group. | From baseline until end of trial at week 48 or 60, depending on the dose group.
Change and percent change compared with pre-dose baseline of platelet inhibition at different time points in each group. | From randomization until week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Ribocure Clinic, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: Undecided